CLINICAL TRIAL: NCT04547751
Title: Hospitalisations of Teenagers and Young Adulthoods in Mayotte After Consumption of an Illegal Drug Called " Chimique ", Which Substances Are Incriminated ? : HOMACHI
Acronym: HOMACHI
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: ARS (Agence Régionale de Santé) Mayotte (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/27
Record Dates: First submitted 2019-10-11; First posted 2020-09-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Drug Abuse
Keywords: drug abuse; chimique; High resolution mass spectrometry
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult: Patients aged 18yrs and older hospitalized in the Emergency Department of the Mayotte Hospital Center after taking a chemical or other psychoactive substance and for whom a blood test is required
  Interventions: Other: targeted high-resolution mass spectrometry
- Minor: Patients aged 14-17yrs and older hospitalized in the Emergency Department of the Mayotte Hospital Center after taking a chemical or other psychoactive substance and for whom a blood test is required
  Interventions: Other: targeted high-resolution mass spectrometry

INTERVENTIONS:
Other: targeted high-resolution mass spectrometry — difference between the number of new substances identified using targeted analysis by liquid chromatography coupled with high-resolution mass spectrometry versus using targeted analysis. "narcotics-new substance" by liquid chromatography coupled with tandem mass spectrometry

SUMMARY:
The study aims (i) to identify which substances leading to hospitalizations at Mayotte are also called "chimique" and (ii) to correlate these substances with clinical pictures in order to favor a better approach of the treatments.

DETAILED DESCRIPTION:
The CEIP-A of Bordeaux (in charge of French overseas departments) has been commissioned by the MILD&CA in 2015 to reinforce the links between local caregivers and the addictoviligance's inquieries. In particular, the CEIP-A has been alerted about a drug called " chimique " in Mayotte, leading to many hospitalizations. Most of the patients are less than 18 year old or are young adulthoods. For all patients who have agreed to participate in this study, the remainder of the blood sample will be reused for a drop of blood on blotting paper; the remainder of the remainder will be stored in the heparinized tube. Medical data collected in the emergency department will also be collected. All the data will be analyzed by the pharmacology and toxicology laboratory of the Bordeaux University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the Emergency Department of the Mayotte Hospital Center after taking a chemical or other psychoactive substance and for whom a blood test is required;
* Age ≥ 14 years.

Exclusion Criteria:

* Patient without parental authority for minor patients aged 14yrs; Patient not included in the exception article 59 of the law of January 6th, 1978 modified for patient aged 15yrs and older

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in the Emergency Department of the Mayotte Hospital Center after taking a chemical or other psychoactive substance
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
number of new substances identified | Baseline
  number of new substances identified

SECONDARY OUTCOMES:
Active ingredients found | Baseline
  Number of active ingredients found (including new substances

CONTACTS AND LOCATIONS:
Locations (1):
- CH Mayotte, Mayotte, France, France

IPD SHARING:
Plan to Share IPD: No